CLINICAL TRIAL: NCT03161808
Title: Rare CFTR Mutation Cell Collection Protocol (RARE)
Acronym: RARE
Status: Recruiting | Type: Observational
Sponsor: George Solomon (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, George Solomon, MD, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Other Study IDs: RARE-OB-16
Record Dates: First submitted 2017-05-09; First posted 2017-05-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal epithelial cells and blood (to confirm CFTR genotype and to derive iPSCs) will be collected from all subjects; consent for whole genome sequencing analysis will be obtained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over 1,900 mutations in the gene for the cystic fibrosis transmembrane conductance regulator (CFTR) protein are implicated in causing Cystic Fibrosis (CF). Potential therapies that directly target defective CFTR are being evaluated in important clinical trials, but most target the most common CFTR mutation F508del. Many patients with rare CF mutations are not able to participate in those studies. The RARE study is specifically designed for people with CF caused by rare mutations. Eligible rare mutations are listed below:

• CF patients who are heterozygous for pre-mature stop codons as noted below: i. one allele must be a F508del ii. the other allele must be a pre-mature stop codon mutation

• CF Patients with other genotypes that require Study PI permission: i. CF patients with two mutations that are not eligible for Trikafta ii. CF patients homozygous or heterozygous (other allele must be F508del) for rare mutations of special interest (e.g., 711+3A->G, 2789+5G->A, 3272-26A->G, 3849+10kbC->T). Other rare mutations will be considered on a case by case basis

This is a multi-site, specimen collection study. Investigators will collect blood, intestinal cells and nasal cells from each participant. Cells from these specimens will be used to test future CFTR modulators to see if they might work for people with study eligible rare mutations. Having cells to test in the lab is an important first step in identifying potential new therapies for people with these mutations.

DETAILED DESCRIPTION:
This is a multi-site, specimen collection study for people with Cystic Fibrosis who have rare mutations. This study is non-interventional so there is no study drug or investigational treatment involved.

* Once a potentially eligible participant is identified (either self-identified or by their CF care center), and the person has expressed interest in participating in the study, the participant will be referred to a participating study site to receive additional information about the study and about travel arrangements (if needed).
* The eligibility criteria are broad and inclusive: Often studies have restrictions around lung function that limit who can participate. The only real restriction for this study rare mutations as defined on the RARE study eligible mutations list.
* Blood, intestinal cells, nasal cells will be collected from all participants.
* Participants will be compensated for the time of the visit and travel expenses will be pre-paid by the study. The study site research coordinator can provide more detail on how much participants will be paid.
* This study is being conducted at six regional sites. Participants may travel to any of the regional study sites to participate, but the participant will need to talk with the research coordinator at the site of their choice to get all of the study details before making a decision to participate. The study site research coordinator will put participants in contact with the travel agency to arrange and pre-pay for travel (including hotel, airline/train arrangements as needed).

Visit Schedule:

Two day study visit

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 12 years of age at time of consent
* Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with CF and one or more of the following criteria (1. Sweat chloride ≥ 60 milliequivalents/Liter (mEq/L) by quantitative pilocarpineiontophoresis test (QPIT) OR upon permission of the RARE Investigator- Sponsors, 2. Two well-characterized mutations in the cystic fibrosis transmembrane conductive regulator (CFTR) gene, 3.Abnormal nasal potential difference (NPD) (change in NPD in response to a low chloride solution and isoproterenol of lessthan -6.6 mV)
* Confirmed genotype of the current recruitment focus for certain target rare mutations. The initial recruitment focus will be CF patients who are homozygous for pre-mature stop codons. Operations Memos will detail any future current genotype targets.
* Written informed consent (and assent when applicable) obtained from participant or participant's legal representative and ability to comply with the requirements of the study.
* Willing to travel (if needed) to a regional study site for cell collection.

Exclusion Criteria:

1. Presence of a medical condition, abnormality, or laboratory value(s) that in the opinion of the onsite principal investigator and/or collaborating gastroenterologist may compromise the quality of the data or place the subject at significant risk by undergoing the research related biopsy, including:

   Significantly diseased distal rectal/GI tissue that could place the participant at risk by participating in the study (as judged by the collaborating gastroenterologist, such as significant hemorrhoids, vascular abnormalities, colonic infection, radiation injury or history of radiation therapy to the rectum, prostate and/or pelvic area)

   Any of the following abnormal lab values at the study visit:

   i. Platelets < 50 x 10^3/µL ii. Hemoglobin < 10 gm/dL iii. Hematocrit < 30% iv. WBC > 20 x 10^3/µL v. Neutropenia (ANC < 1.5 x 10^3/µL) vi. Lymphopenia (absolute lymphocyte count < 1.5 x 10^3/µL) vii. PT/INR > 1.5 viii. Other bleeding diathesis
2. Positive pregnancy test (for female of childbearing potential) at the study visit.
3. Breastfeeding (if patient opts to use sedation).
4. Current use of drugs with significant risks of compromising immunity (e.g. oral steroid use >20 mg/day) for >14 days prior to the rectal biopsy.
5. History of organ transplant.
6. Use of oral anticoagulant medications (e.g., chronic anticoagulant therapy such as warfarin or platelet inactivators such as aspirin) within seven days prior to rectal biopsy.
7. Unable or unwilling to withhold use of oral anticoagulant medications (e.g., chronic anticoagulant therapy such as warfarin or platelet inactivators such as aspirin) within 7 days after rectal biopsy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a diagnosis of CF who meet all of the inclusion and none of the exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The Number of samples collected from cystic fibrosis participants with rare CFTR mutations | 2-5 year observational period
  CFTR mutations will be confirmed. Once the mutations are confirmed as RARE study eligible mutations, the specimen(s) collected will be expanded, added to a specimen bank and made available to the research community for the evaluation of potential CFTR modulating agents.
The number of nasal cells collected | 2-5 year observational period
  Nasal cells will be collected from all participants.
Number of Blood samples | 2-5 year observational period
  Blood samples will be collected from all participants
Number of rectal samples collected | 2-5 year observational period
  Rectal biopsy samples will be collected from all participants

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No